CLINICAL TRIAL: NCT00014391
Title: A Randomized Double-Blind Placebo-Controlled Phase III Study To Evaluate The Safety And Efficacy Of Palivizumab Combined With Aerosolized Ribavirin Compared To Ribavirin Alone To Treat RSV Pneumonia In Patients With Bone Marrow Transplants (BMT)
Brief Title: Ribavirin With or Without Monoclonal Antibody Therapy in Treating Patients Who Develop RSV Pneumonia Following Peripheral Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: 1379.00; FHCRC-1379.00; NCI-G01-1929; CDR0000068540 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-04-10; First posted 2004-04-13 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; recurrent childhood rhabdomyosarcoma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; chronic idiopathic myelofibrosis; childhood acute promyelocytic leukemia (M3); testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; refractory hairy cell leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent ovarian germ cell tumor; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; infection; pulmonary complications; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; previously treated childhood rhabdomyosarcoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Infections; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Palivizumab; Ribavirin

INTERVENTIONS:
Biological: palivizumab
Drug: ribavirin

SUMMARY:
RATIONALE: Antivirals such as ribavirin are used to treat infections caused by viruses. It is not yet known if ribavirin is more effective with or without monoclonal antibody therapy in treating patients who develop RSV pneumonia following peripheral stem cell transplantation.

PURPOSE: Randomized phase III trial to compare the effectiveness of ribavirin with or without monoclonal antibody in treating patients who develop RSV pneumonia following peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy, in terms of all-cause mortality reduction, of ribavirin with or without palivizumab in patients with respiratory syncytial virus pneumonia following stem cell transplantation. II. Determine the safety of these treatments in this patient population.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to prior ribavirin exposure for this infection (24 hours or more vs less than 24 hours) and requirement for ventilator support (yes vs no). Patients are randomized to one of two treatment arms. Arm I: Patients receive aerosolized ribavirin via face mask or oxygen tent over 2 hours 3 times daily or over 16-18 hours on days 1-10 and palivizumab IV 2 hours before ribavirin administration on day 1. Arm II: Patients receive aerosolized ribavirin as in arm I and placebo IV 2 hours before ribavirin administration on day 1. Patients are followed at 14, 21, and 28 days.

PROJECTED ACCRUAL: A total of 140 patients (70 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Confirmed respiratory syncytial virus (RSV) pneumonia documented by rapid antigen test (ELISA or IFA), shell vial culture of bronchoalveolar lavage specimens, or tissue antigen staining of lung biopsy sample New infiltrate on chest x-ray and at least one of the following: Cough Wheezing Dyspnea and/or tachypnea (greater than 150% of baseline) Oxygen saturation less than 90% on two occasions 1 hour apart on room air Arterial oxygen pressure less than 80 No more than 60 hours since confirmation of pneumonia by chest x-ray Received prior stem cell transplantation and meet one of the following: Between start of conditioning (preparative) regimen and day 90 after allogeneic, autologous, or syngeneic stem cell transplantation (SCT) Between days 91 and 180 after unrelated HLA mismatch-related allogeneic SCT (bone marrow, peripheral blood stem cells (PBSC), or cord blood), T-cell depleted allogeneic transplantation, or CD34 selected allogeneic PBSC transplantation Between days 91 and 180 after SCT with graft-versus-host disease requiring systemic steroids expected to continue throughout study Other pulmonary pathogens in addition to RSV allowed

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: At least 48 hours Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No prior adverse reaction to ribavirin or palivizumab No allergy to monoclonal antibodies HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 3 months since prior immunotherapy for respiratory syncytial virus (RSV) including RSV hyperimmune globulin or other RSV monoclonal antibodies Concurrent IV immunoglobulin allowed No prior experimental RSV vaccine No concurrent RSV hyperimmune globulin No other concurrent RSV-specific monoclonal antibodies Chemotherapy: Not specified Endocrine therapy: See Disease Characteristics Radiotherapy: Not specified Surgery: Not specified Other: At least 4 weeks since prior investigational products for respiratory viral diseases At least 3 months since prior anti-viral drugs with specific anti-RSV activity Prior aerosolized ribavirin allowed No other concurrent anti-viral drugs with specific anti-RSV activity Concurrent ganciclovir or foscarnet allowed Ventilator support allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-02; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States